CLINICAL TRIAL: NCT00005166
Title: Sodium Transport: Genetics and Hypertension
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1040; R01HL030428 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
Originally, to determine whether genetic alterations in pathways of sodium ion transport in the red blood cells of children could predict their risk of developing primary hypertension in adulthood. In 1992, the objective was to determine the genetic basis of interindividual variation in the risk of essential hypertension in the population at large using the Rochester Family Heart Study.

DETAILED DESCRIPTION:
BACKGROUND:

Blood pressure has a continuous unimodal distribution in the general population. Individuals with levels elevated above the 80th percentile suffer from hypertension, a major cause of cardiovascular morbidity and mortality. Over 95 percent of hypertensives have no other primary disease and are said to have essential hypertension. Pedigree and twin studies indicate that genetic differences account for a large fraction of the interindividual variation in blood pressure. In 1984 when the study began, no genetic loci had yet been identified that were useful markers for essential hypertension or served as probes into the biological basis for interindividual blood pressure variability. Environmental factors also influence blood pressure; increased dietary intake of sodium chloride, in particular, elevates blood pressure and may contribute to the development of essential hypertension in some people. It was hypothesized that genetically determined alterations in the metabolism of sodium ion occur in a subset of the population that is at increased liability to develop elevated blood pressure upon exposure to the usual range of dietary sodium intake

Reports of altered sodium transport in the red blood cells of individuals with essential hypertension and their offspring stimulated interest in this hypothesis. Several proposals were offered to explain how alterations in sodium transport similar to those observed in red blood cells could lead to elevated blood pressure when present in the renal tubules or vascular smooth muscle. Studies of the sodium-lithium countertransport system indicated that red blood cell sodium transport pathways may provide informative phenotypes that relate blood pressure and essential hypertension more closely with genetic factors.

Numerous laboratories have confirmed that the maximal rate of sodium-lithium countertransport is increased in red blood cells from individuals with essential hypertension. The sodium-lithium countertransport is normal in secondary forms of hypertension and increased levels in essential hypertension cannot be attributed to age, body size, gender or dietary salt intake. The highest levels are observed in individuals with a positive family history of essential hypertension and the lowest levels occur in normotensive controls without hypertensive relatives.

DESIGN NARRATIVE:

When the study began in 1984, the objective was to determine whether genetic alterations in pathways of sodium transport in the red blood cells of children could predict their risk of developing primary hypertension in adulthood. Approximately 600 children between 7 and 18 years of age were randomly selected as index cases for family studies. Each participating member of the pedigrees studied underwent venipuncture for withdrawal of whole blood. A medical history was obtained from each family member visiting the clinic and a physical examination was conducted. Existing medical records for all living and deceased adult relatives in the 600 pedigrees were reviewed. In addition, 40 normotensive adult members of 300 pedigrees underwent metabolic balance and renal clearance studies, as well as ambulatory blood pressure recordings. Segregation analysis of pedigree data was carried out to determine the most likely mode for genetic transmission of the sodium-lithium counter-transport phenotype. Baseline genetic information about sodium-lithium was related to the prevalence of primary hypertension in the families of index children. Additional phenotypes involved in blood pressure regulation were also studied including renal proximal tubular sodium reabsorption, atrial natriuretic peptide, sodium-potassium adenosinetriphosphate pump, and sodium-potassium cotransport.

The study was renewed several times, the last in 1992 to continue work on the genetic basis of interindividual variation in risk of essential hypertension in the population at large using the Rochester Family Heart Study (RFHS). The RFHS was used to address three major questions: 1) Which intermediate biochemical, physiological, and anthropomorphic traits predicted blood pressure and contributed to the pathogenesis of essential hypertension 2) Did allelic variation in one or more genes have large effects on any of these intermediate traits? 3) Did information about allelic variation improve prediction of risk of essential hypertension beyond what was provided by measure of the intermediate traits?

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1984-04; Study Completion 1996-03 (Actual)

REFERENCES:
- [Background] Boerwinkle E, Turner ST, Sing CF. The role of the genetics of sodium lithium countertransport in the determination of blood pressure variability in the population at large. Prog Clin Biol Res. 1984;165:479-507. No abstract available. PMID 6504919
- [Background] Sing CF, Boerwinkle E: The Genetics of Blood Pressure Variability: An Overview. In: Proceedings, Children's Blood Pressure: The Eighty-Eighth Ross Conference on Pediatric Research. Ross Laboratories, 1984
- [Background] Turner ST, Fairbanks VF. Is measurement of erythrocyte Na+ influx useful for ascertainment of essential hypertension? Mayo Clin Proc. 1984 Jul;59(7):506-8. doi: 10.1016/s0025-6196(12)60442-x. No abstract available. PMID 6738116
- [Background] Turner ST, Johnson M, Boerwinkle E, Richelson E, Taswell HF, Sing CF. Sodium-lithium countertransport and blood pressure in healthy blood donors. Hypertension. 1985 Nov-Dec;7(6 Pt 1):955-62. doi: 10.1161/01.hyp.7.6.955. PMID 4077225
- [Background] Boerwinkle E, Chakraborty R, Sing CF. The use of measured genotype information in the analysis of quantitative phenotypes in man. I. Models and analytical methods. Ann Hum Genet. 1986 May;50(2):181-94. doi: 10.1111/j.1469-1809.1986.tb01037.x. PMID 3435047
- [Background] Sing CF, Boerwinkle E, Turner ST. Genetics of primary hypertension. Clin Exp Hypertens A. 1986;8(4-5):623-51. doi: 10.3109/10641968609046580. PMID 3530548
- [Background] Richelson E, Snyder K, Carlson J, Johnson M, Turner S, Lumry A, Boerwinkle E, Sing CF. Lithium ion transport by erythrocytes of randomly selected blood donors and manic-depressive patients: lack of association with affective illness. Am J Psychiatry. 1986 Apr;143(4):457-62. doi: 10.1176/ajp.143.4.457. PMID 2420218
- [Background] Boerwinkle E, Turner ST, Weinshilboum R, Johnson M, Richelson E, Sing CF. Analysis of the distribution of erythrocyte sodium lithium countertransport in a sample representative of the general population. Genet Epidemiol. 1986;3(5):365-78. doi: 10.1002/gepi.1370030509. PMID 3781241
- [Background] Turner ST, Boerwinkle E, Johnson M, Richelson E, Sing CF. Sodium-lithium countertransport in ambulatory hypertensive and normotensive patients. Hypertension. 1987 Jan;9(1):24-34. doi: 10.1161/01.hyp.9.1.24. PMID 2432010
- [Background] Turner ST, Weidman WH, Michels VV, Reed TJ, Ormson CL, Fuller T, Sing CF. Distribution of sodium-lithium countertransport and blood pressure in Caucasians five to eighty-nine years of age. Hypertension. 1989 Apr;13(4):378-91. doi: 10.1161/01.hyp.13.4.378. PMID 2925236
- [Background] Rebbeck TR, Turner ST, Michels VV, Moll PP. Genetic and environmental explanations for the distribution of sodium-lithium countertransport in pedigrees from Rochester, MN. Am J Hum Genet. 1991 Jun;48(6):1092-104. PMID 2035530
- [Background] Sing CF, Haviland MB, Templeton AR, Zerba KE, Reilly SL. Biological complexity and strategies for finding DNA variations responsible for inter-individual variation in risk of a common chronic disease, coronary artery disease. Ann Med. 1992 Dec;24(6):539-47. doi: 10.3109/07853899209167008. PMID 1485951
- [Background] Reilly SL, Ferrell RE, Kottke BA, Sing CF. The gender-specific apolipoprotein E genotype influence on the distribution of plasma lipids and apolipoproteins in the population of Rochester, Minnesota. II. Regression relationships with concomitants. Am J Hum Genet. 1992 Dec;51(6):1311-24. PMID 1463013
- [Background] Turner ST, Rebbeck TR, Sing CF. Sodium-lithium countertransport and probability of hypertension in Caucasians 47 to 89 years old. Hypertension. 1992 Dec;20(6):841-50. doi: 10.1161/01.hyp.20.6.841. PMID 1452301
- [Background] Schwartz GL, Turner ST, Sing CF. Twenty-four-hour blood pressure profiles in normotensive sons of hypertensive parents. Hypertension. 1992 Dec;20(6):834-40. doi: 10.1161/01.hyp.20.6.834. PMID 1452300
- [Background] Mailly F, Moll P, Kottke BA, Kamboh MI, Humphries SE, Ferrell RE. Estimation of the frequency of isoform-genotype discrepancies at the apolipoprotein E locus in heterozygotes for the isoforms. Genet Epidemiol. 1992;9(4):239-48. doi: 10.1002/gepi.1370090403. PMID 1398044
- [Background] Reilly SL, Ferrell RE, Kottke BA, Kamboh MI, Sing CF. The gender-specific apolipoprotein E genotype influence on the distribution of lipids and apolipoproteins in the population of Rochester, MN. I. Pleiotropic effects on means and variances. Am J Hum Genet. 1991 Dec;49(6):1155-66. PMID 1842218
- [Background] Kottke BA, Moll PP, Michels VV, Weidman WH. Levels of lipids, lipoproteins, and apolipoproteins in a defined population. Mayo Clin Proc. 1991 Dec;66(12):1198-208. doi: 10.1016/s0025-6196(12)62470-7. PMID 1749288
- [Background] Kaprio J, Ferrell RE, Kottke BA, Kamboh MI, Sing CF. Effects of polymorphisms in apolipoproteins E, A-IV, and H on quantitative traits related to risk for cardiovascular disease. Arterioscler Thromb. 1991 Sep-Oct;11(5):1330-48. doi: 10.1161/01.atv.11.5.1330. PMID 1911720
- [Background] Turner ST, Michels VV. Sodium-lithium countertransport and hypertension in Rochester, Minnesota. Hypertension. 1991 Aug;18(2):183-90. doi: 10.1161/01.hyp.18.2.183. PMID 1885226
- [Background] Perusse L, Moll PP, Sing CF. Evidence that a single gene with gender- and age-dependent effects influences systolic blood pressure determination in a population-based sample. Am J Hum Genet. 1991 Jul;49(1):94-105. PMID 2063879
- [Background] Reilly SL, Kottke BA, Sing CF. The effects of generation and gender on the joint distributions of lipid and apolipoprotein phenotypes in the population at large. J Clin Epidemiol. 1990;43(9):921-40. doi: 10.1016/0895-4356(90)90076-2. PMID 2213081
- [Background] Kwon JM, Boehnke M, Burns TL, Moll PP. Commingling and segregation analyses: comparison of results from a simulation study of a quantitative trait. Genet Epidemiol. 1990;7(1):57-68. doi: 10.1002/gepi.1370070113. PMID 2184092
- [Background] Zerba KE, Friedlaender JS, Sing CF. Heterogeneity of the blood pressure distribution among Solomon Islands societies with increasing acculturation. Am J Phys Anthropol. 1990 Apr;81(4):493-511. doi: 10.1002/ajpa.1330810406. PMID 2333938
- [Background] Rebbeck TR, Turner ST, Sing CF. Sodium-lithium countertransport genotype and the probability of hypertension in adults. Hypertension. 1993 Oct;22(4):560-8. doi: 10.1161/01.hyp.22.4.560. PMID 8406661
- [Background] Reilly SL, Sing CF, Savageau MA, Turner ST. Analysis of systems influencing renal hemodynamics and sodium excretion. I. Biochemical systems theory. Integr Physiol Behav Sci. 1994 Jan-Mar;29(1):55-73. doi: 10.1007/BF02691281. PMID 8018552
- [Background] Turner ST, Reilly SL. Renal sodium excretion in sons of hypertensive parents. Hypertension. 1993 Sep;22(3):323-30. doi: 10.1161/01.hyp.22.3.323. PMID 8349325
- [Background] Kardia SL, Sing CF, Turner ST. The response of renal plasma flow to angiotensin II infusion in a population-based sample and its association with the parental history of essential hypertension. J Hypertens. 1997 May;15(5):483-93. doi: 10.1097/00004872-199715050-00003. PMID 9170000
- [Background] Stengard JH, Zerba KE, Turner ST, Sing CF. A biometrical study of the relationship between sodium-lithium countertransport and triglycerides. Ann Hum Genet. 1997 Mar;61(Pt 2):121-36. doi: 10.1046/j.1469-1809.1997.6120121.x. PMID 9177119
- [Background] Turner ST, Sing CF. Erythrocyte sodium transport and the probability of having hypertension. J Hypertens. 1996 Jul;14(7):829-37. doi: 10.1097/00004872-199607000-00005. PMID 8818921
- [Background] Flickinger AL, Lerman LO, Sheedy PF 2nd, Turner ST. The relationship between renal cortical volume and predisposition to hypertension. Am J Hypertens. 1996 Aug;9(8):779-86. doi: 10.1016/0895-7061(96)00097-0. PMID 8862224
- [Background] Schwartz GL, Turner ST, Sing CF. Association of genetic variation with interindividual variation in ambulatory blood pressure. J Hypertens. 1996 Feb;14(2):251-8. doi: 10.1097/00004872-199602000-00015. PMID 8728304
- [Background] Rebbeck TR, Turner ST, Sing CF. Probability of having hypertension: effects of sex, history of hypertension in parents, and other risk factors. J Clin Epidemiol. 1996 Jul;49(7):727-34. doi: 10.1016/0895-4356(96)00015-7. PMID 8691221
- [Background] Flickinger AL, Burnett JC Jr, Turner ST. Atrial natriuretic peptide and blood pressure in a population-based sample. Mayo Clin Proc. 1995 Oct;70(10):932-8. doi: 10.4065/70.10.932. PMID 7564543
- [Background] Turner ST, Reilly SL. Fallacy of indexing renal and systemic hemodynamic measurements for body surface area. Am J Physiol. 1995 Apr;268(4 Pt 2):R978-88. doi: 10.1152/ajpregu.1995.268.4.R978. PMID 7733408
- [Background] Sing CF, Moll PP. Genetics of atherosclerosis. Annu Rev Genet. 1990;24:171-87. doi: 10.1146/annurev.ge.24.120190.001131. No abstract available. PMID 2088166